CLINICAL TRIAL: NCT03031457
Title: Microsurgical Breast Reconstruction - Identifying Procedure-Specific Risk Factors for Venous Thromboembolism
Brief Title: Microsurgical Breast Reconstruction & VTE
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Arash Momeni, Assistant Professor of Surgery, Stanford University
Other Study IDs: 39855
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Breast Reconstruction; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients undergo primary fascial closure of abdominal donor-site
  Interventions: Diagnostic Test: Duplex ultrasound

INTERVENTIONS:
Diagnostic Test: Duplex ultrasound — Duplex ultrasound of lower extremity venous system

SUMMARY:
Venous thromboembolism (VTE) encompasses pulmonary embolism (PE) and deep venous thrombosis (DVT) and continues to be a major patient safety issue after reconstructive plastic surgery. Significant morbidity and mortality is associated with VTE events. This disease entity represents the most common cause of preventable in-hospital death as evidenced by over 100,000 annual VTE-related deaths in the U.S. The associated economic burden is substantial, with annual costs to the U.S. healthcare system in excess of $7 billion.

Cancer patients have been identified as a particularly vulnerable patient population. Of these, breast cancer patients represent the largest group treated by plastic surgeons. An increasing number of breast reconstructions are performed in the U.S. with a documented 35% increase in the annual number of breast reconstructions since 2000. Over 106,000 breast reconstructions were performed in 2015 alone.

Of all reconstructive modalities, autologous breast reconstruction using abdominal flaps is associated with the highest risk for VTE. We believe that a key element rendering these patients susceptible to postoperative VTE is inadequate duration of chemoprophylaxis. This is supported by the observation that VTE risk remains elevated for up to 12 weeks postoperatively. We hypothesize that lower extremity deep venous system stasis is a procedure-specific key contributing factor to postoperative VTE risk.

This study examines the duration of postoperative lower extremity venous stasis to identify patients who might benefit from extended chemoprophylaxis. We will use Duplex imaging technology to examine the lower extremity deep venous system preoperatively, on postoperative day 1, and on the day of discharge to determine if patients display radiographic evidence of lower extremity venous stasis at the time of hospital discharge.

A better understanding of pathophysiologic mechanisms that contribute to the development of VTE as well as surgical means that reduce VTE risk factors have the potential to optimize VTE prophylaxis, thus, favorably impacting clinical outcome in a large patient population.

ELIGIBILITY:
Inclusion Criteria:

* see study population description

Exclusion Criteria:

* Superficial inferior epigastric artery flaps
* Donor-sites other than the abdomen
* Chronic obstructive pulmonary disease (COPD)
* Liver disease.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Adult (age ≥18 years) female patients who are scheduled to undergo autologous breast reconstruction following mastectomy. Only patients who undergo breast reconstruction with free abdominal flaps that require violation of the anterior rectus sheath, i.e. MS-TRAM and DIEP flaps, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Vessel diameter (in cm) | 1 Day of discharge
Cross-sectional area (in cm^2) | 1 Day of discharge
Flow velocity (in cm/sec) | 1 Day of discharge

SECONDARY OUTCOMES:
90-day VTE event | 90-day
Abdominal hernia/bulge rate at 1 year postop | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arash Momeni, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Momeni A, Sorice SC, Li AY, Nguyen DH, Pannucci C. Breast Reconstruction with Free Abdominal Flaps Is Associated with Persistent Lower Extremity Venous Stasis. Plast Reconstr Surg. 2019 Jun;143(6):1144e-1150e. doi: 10.1097/PRS.0000000000005613. PMID 30907811